CLINICAL TRIAL: NCT06550791
Title: A Prospective Feasibility Study Evaluating the Implementation of the Anticancer Lifestyle Program in Endometrial Cancer Survivors
Brief Title: Evaluating the Anticancer Learning Circle Lifestyle Program in Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kari Ring, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR230435
Record Dates: First submitted 2024-07-29; First posted 2024-08-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Neoplasm, Uterine
Keywords: Endometrial Cancer; Holistic Cancer Treatment; Lifestyle Change
MeSH Terms: conditions — Uterine Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anticancer Learning Circle Participant (Experimental)
  Interventions: Behavioral: Anticancer Learning Circle

INTERVENTIONS:
Behavioral: Anticancer Learning Circle — All participants will partake in the Anticancer Learning Circle, a lifestyle modification program. All participants will complete web-based learning modules focused on improving diet, lowering stress, increasing fitness, and reducing exposure to toxins in the home environment. Each week, all participants will meet as a group to discuss the learning topic of the web-based learning module for the week.

SUMMARY:
The purpose of this study is to promote positive lifestyle change among endometrial cancer survivors by using a group-based intervention. Endometrial cancer survivors are at an increased risk of other health conditions like heart disease, diabetes, and other cancers. The study team at the University of Virginia wants to explore new ways to lower these risks. This study will be evaluating the Anticancer Lifestyle program, which takes a more holistic approach and uses web-based learning modules along with weekly group sessions to discuss each topic of the web-based learning modules.

ELIGIBILITY:
Inclusion Criteria:

* History of stage I-IV endometrial cancer, any histologic subtype
* Completed cancer treatment, and in surveillance
* Have no evidence of endometrial cancer as determined by primary oncologist
* Be at least 18 years of age
* Be able to read and communicate in English
* Have a smartphone with access to cellular service or computer access with internet service
* Must have technological competency/proficiency to use their Smartphone and/or computer, as self-reported by potential subject
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Pregnant women
* Prisoners
* Subject is blind

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Person born with a uterus
Enrollment: 23 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Number of participants that complete the program | Week 7
  The proportion of participants completing the program as defined by the number of those who participated in at least 75% of online sessions.

SECONDARY OUTCOMES:
Change from Week 0 of the Automated Self-administered 24-hour Dietary Assessment (ASA24) at Week 7 | 7 weeks
  The Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool is a free, web-based tool created by the National Cancer Institute to assess nutritional intake. ASA24 enables multiple, automatically coded, self-administered 24-hour diet recalls and/or single or multi-day food records, also known as food diaries.
  Overall nutrition will be assessed at week 0 and week 7 to compare and evaluate changes in dietary patterns of participants.
Change from Week 0 of Generalized Anxiety Disorder (GAD-7) Survey from Baseline at Week 32 | 32 weeks
  The GAD-7 is a validated, self-reported survey assessing feelings of anxiety. Possible scores range from 0 (minimal anxiety) to 21 (severe anxiety).
  Scores will be evaluated at weeks 0, 4, 7, and 32 with overall primary endpoint evaluating change between week 0 and week 32.
  Change = (Week 32 Score - Week 0 score)
Change from Week 0 of the Godin Leisure-Time Exercise Questionnaire (GLTEQ) from Baseline at Week 32 | 32 weeks
  The GLTEQ is a validated, self-reported scale assessing physical activity. Participants self-report the number of times per week they engage in strenuous, moderate, and mild/light physical activity. The self-reported number is multiplied by 9 for strenuous exercise, 5 for moderate exercise, and 3 for mild/light exercise. Scores can range from less than 14 units (insufficiently Active/Sedentary) to 24 units of more (Active).
  Scores will be evaluated at weeks 0, 4, 7, and 32 with overall primary endpoint evaluating change between week 0 and week 32.
  Change = (Week 32 score - Week 0 score)
Change from Week 0 of the Cancer Worry Scale (CWS) to Week 32 | 32 weeks
  The CWS scale is a validated, self-reported scale assessing participants worries about developing or reoccurring cancer. Scores can range from 8 (seldom or never worried) to 32 (worried a lot/almost all the time).
  Scores will be evaluated at weeks 0, 4, 7, and 32 with overall primary endpoint evaluating change between week 0 and week 32.
  Change = (Week 32 score - Week 0 score)
Change from Week 0 of the Patient Health Questionnaire (PHQ-9) to Week 32 | Baseline and Week 32
  The PHQ-9 is a validated, self-reported scale to assess symptoms of major depressive disorder. Scores can range from 0 (none-Minimal) to 27 (severe).
  Scores will be evaluated at weeks 0, 4, 7, and 32 with overall primary endpoint evaluating change between week 0 and week 32.
  Change = (Week 32 score - Week 0 score)
Assess Attitudes Toward Group-Based Lifestyle Therapy Program Utilizing Internal Scale at Week 7 and Week 32 | Week 7 and Week 32
  Internal survey built to evaluate participants' satisfaction with the Anticancer Lifestyle Foundation's lifestyle program.
  Quantitative measures are gathered utilizing a scale of Strongly Disagree to Strongly Agree to assess participant attitudes towards program satisfaction, usefulness of information learned, and to gauge if the participant feels they were able to make positive lifestyle changes through participation in the program.
  Additional questions assess feelings towards preferences of group size, platform used, number of sessions, and length of program.
  Qualitive measure allows participants to share any thoughts/concerns/or feedback regarding the program.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Ring, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No